CLINICAL TRIAL: NCT06335901
Title: Clinical Characteristics and Outcomes of Coronary Heart Disease: a Prospective Cohort Study
Brief Title: Clinical Characteristics and Outcomes of Coronary Heart Disease
Acronym: IMPROVE
Status: Completed | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Xiangxie, MD,The First Affiliated Hospital Of XinJiang Medicial University, Xinjiang Medical University
Other Study IDs: xx20190901
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 2
  Interventions: Drug: Drug:Standard therapy

INTERVENTIONS:
Drug: Drug:Standard therapy — Percutaneous coronary Intervention

SUMMARY:
This study evaluated and compared the prognostic value of different Baseline data and clinical variables to develop predictive model in patients with CHD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Coronary Heart Disease (CHD) admitted to the First Affiliated Hospital of Xinjiang Medical University.
2. The diagnosis is based on clinical assessments, including symptomatic evaluation, electrocardiographic findings, and coronary angiography.

Exclusion Criteria:

We excluded patients who had serious heart failure, malignant tumor，rheumatic heart disease, valvular heart disease, congenital heart disease, pulmonary heart disease and serious dysfunction of the liver or kidney.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease hospitalized at the First Affiliated Hospital of Xinjiang Medical University.
Sampling Method: Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Death （All-cause mortality、Cardiac mortality ） | 5 years of follow-up deaths occurred during this period

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 5 years of follow-up deaths occurred during this period

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No